CLINICAL TRIAL: NCT04006899
Title: Development of a Segmental Bioelectrical Impedance Spectroscopy Device for Body Composition Measurement
Status: Completed | Type: Observational
Sponsor: Jun Choi (Other)
Responsible Party: Sponsor-Investigator, Jun Choi, Assistant Professor, Georgia Southern University
Organization: Georgia Southern University (Other)
Other Study IDs: GSU001
Record Dates: First submitted 2019-06-28; First posted 2019-07-05 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Medical Device
Keywords: Bioelectrical Impedance spectroscopy; Body compositions; Segmental Bioelectrical impedance spectroscopy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- subj 1: Three commercially available BIA devices vs SBIS device
  Interventions: Device: Bioelectrical Impedance Monitor

INTERVENTIONS:
Device: Bioelectrical Impedance Monitor — Subjects had been under the test of three commercially available devices and the device that the investigators had developed.

SUMMARY:
A device for measuring body composition with a small electric current, at 200 μA, (bioelectrical impedance analysis, or BIA) was designed. The goal of this study is to validate the device against several existing devices using the same method of measuring body composition with a small electric current.

DETAILED DESCRIPTION:
The measurement of individual segments, instead of the body as a whole, with BIA has not been fully explored. The prototype device is capable of directly measuring multiple body segments (arm, trunk, and leg) simultaneously, and the final version will be able to provide composition about each segment and the body as a whole. Current devices on the market are not capable of this.

The reference devices will be used to measure segments as well, and the raw measurements will be compared. The Multiscan 5000 provides segmental body composition for the arm or leg, but requires measuring it separately. The SFB7 is designed only for measuring the whole body, but the raw impedance measurement data from the SFB7 can be used for comparison, as the impedance magnitudes of individual segments will be within its measurement range. The Seca 514 doesn't directly measure segments, but it can provide segmental data by measuring from hand to foot, then from hand to hand, and finally from foot to foot. It then uses these measurements, and assumptions about the subject to provide segmental composition data.

ELIGIBILITY:
Inclusion Criteria:

* Students from Georgia Southern University

Exclusion Criteria:

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Students from Georgia Southern University
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2018-06-20 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
Impedance values from each devices | One year IRB period
  Bioelectrical impedance values from three devices were measured and recorded.

CONTACTS AND LOCATIONS:
Overall Officials: junghun choi, Ph.D., Principal Investigator — Georgia Southern University
Locations (1):
- Georgia Southern University, Statesboro, Georgia, United States

IPD SHARING:
Plan to Share IPD: No